CLINICAL TRIAL: NCT05967195
Title: Financial Incentives to Increase Treatment Attendance in First-Episode Psychosis Care: A Non-Randomized, Adaptive Pilot Study
Brief Title: Trial to Increase FEP Attendance
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Penn Innovation in Suicide Prevention for Implementation Research (INSPIRE) Center (Unknown)
Responsible Party: Principal Investigator, William Smith, Principal Investigator, University of Pennsylvania
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-03
Record Dates: First submitted 2023-06-20; First posted 2023-08-01 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-03

CONDITIONS: First-Episode Psychosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Financial Incentive and Text-Messages — Patient-participants will receive modest financial incentive for attending therapy or medication management appointments combined with text messages to encourage attendance at these appointments. Text messages will be informed by principles of behavioral economics. Maximum incentive = $50/month if all appointments attended. Incentives will be pro-rated by percentage of appointments attended. Pro-rating strategies (e.g., uniform amount per appointment, escalating [aka, 'back-loaded'], or decreasing [aka 'frontloaded'] will be sequentially changed based on acceptability and other intervention-related data gathered from participants during the trial.
  Clinician-participants will not receive any intervention, but will receive surveys and interviews to assess their perceptions about the optimization, acceptability, scalability, and other implementation barriers/facilitators for the intervention.

SUMMARY:
Individuals with first-episode psychosis (FEP) are at high-risk for several poor functional and clinical outcomes, including suicide. Coordinated Specialty Care (CSC) is a multidisciplinary, team-based intervention known to improve such outcomes, including suicide risk. However, 30-50% of patients disengage from CSC, thereby limiting its impact. This pilot study will develop and test feasibility of a behavioral change program that uses moderate financial incentives to encourage treatment engagement in 2 CSC programs. A single-arm of 80 patient-participants at these two clinics will be recruited to assess feasibility and acceptability from patient perspectives. Additionally,15 clinicians at these two clinics will be recruited to assess feasibility and acceptability from clinician perspectives, and 50 clinicians from peer clinics not involved in the intervention will be recruited to assess scalability of the intervention. The trial will feature an three-month period for recruitment and baseline data collection and will subsequently feature three intervention periods (3 months each) where modifications to the interventions will be tested (each informed by the feasibility and acceptability findings of the prior period) with the aim of sequentially improving it.

ELIGIBILITY:
Inclusion Criteria:

1. For all participants, age ≥ 18 years old.
2. For intervention trial and patient feasibility and acceptability measurement: Patients with first-episode psychosis, enrolled in Coordinated Specialty Care at the Psychosis Education, Assessment, Care and Empowerment (PEACE) clinic and Psychosis Evaluation and Recovery Center (PERC).
3. For clinician feasibility and acceptability measurement at intervention sites: Clinicians working at PEACE and PERC where the intervention will be piloted.
4. For clinician implementation facilitator and barrier assessment at other Connection LHS sites to assess for scalability: Clinicians in Connection LHS who work at sites other than PEACE and PERC.Participants must sign the informed consent form

Exclusion Criteria:

1. For intervention trial and patient feasibility and acceptability measurement: Expectation of leaving coordinated specialty care programing within 6 months (which will exclude all of the PI's patient panel) and/or intellectual disability of sufficient degree that the patient's primary psychiatrist expects to compromise capacity to consent to this research and/or psychosis secondary to another medical condition (which may not share the same motivational features that are otherwise understood about the primary psychiatric conditions with psychosis).
2. For clinician feasibility and acceptability measurement at intervention sites: Study investigators who work at these clinics will be excluded from participation in the feasibility and acceptability study component given their role in the trial planning and execution.
3. For clinician implementation facilitator and barrier assessment at other Connection LHS sites to assess for scalability: none.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of intervention measure (AIM) | Change at 8 months
  The AIM is a 4-item scale measuring acceptability. Each item is scored 1-5 with 5 indicating greater acceptability. Minimum score is 4; maximum is 20.
Acceptability of intervention measure (AIM) | Change at 6 months
  The AIM is a 4-item scale measuring acceptability. Each item is scored 1-5 with 5 indicating greater acceptability. Minimum score is 4; maximum is 20.
Acceptability of intervention measure (AIM) | Change at 4 months
  The AIM is a 4-item scale measuring acceptability. Each item is scored 1-5 with 5 indicating greater acceptability. Minimum score is 4; maximum is 20.
Feasibility of intervention measure (FIM) | Change at 8 months
  The FIM is a 4-item scale measuring feasibility. Each item is scored 1-5 with 5 indicating greater feasibility. Minimum score is 4; maximum is 20.
Feasibility of intervention measure (FIM) | Change at 6 months
  The FIM is a 4-item scale measuring feasibility. Each item is scored 1-5 with 5 indicating greater feasibility. Minimum score is 4; maximum is 20.
Feasibility of intervention measure (FIM) | Change at 4 months
  The FIM is a 4-item scale measuring feasibility. Each item is scored 1-5 with 5 indicating greater feasibility. Minimum score is 4; maximum is 20.

SECONDARY OUTCOMES:
Implementation Survey Response | Change at 8 months
  Implementation survey. Results will be used to optimize intervention from implementation perspective.
Implementation Survey Response | Change at 6 months
  Implementation survey. Results will be used to optimize intervention from implementation perspective.
Implementation Survey Response | Change at 4 months
  Implementation survey. Results will be used to optimize intervention from implementation perspective.
Motivation Survey Response | Change at 8 months
  Motivation survey. Results will be used to optimize intervention from motivation perspective.
Motivation Survey Response | Change at 6 months
  Motivation survey. Results will be used to optimize intervention from motivation perspective.
Motivation Survey Response | Change at 4 months
  Motivation survey. Results will be used to optimize intervention from motivation perspective.
Ethical Concern Survey Response | Change at 8 months
  Ethical concern survey. Results will be used to optimize intervention from ethical acceptability perspective.
Ethical Concern Survey Response | Change at 6 months
  Ethical concern survey. Results will be used to optimize intervention from ethical acceptability perspective.
Ethical Concern Survey Response | Change at 4 months
  Ethical concern survey. Results will be used to optimize intervention from ethical acceptability perspective.

OTHER OUTCOMES:
attrition | Change at 8 months
  rate of attrition
attrition | Change at 6 months
  rate of attrition
attrition | Change at 4 months
  rate of attrition
psychotic symptomology | Change at 8 months
  Compass-10. The Compass-10 is a self-report scale that measures multiple symptoms associated with psychosis, including mood symptoms. It consists of 10-items, each scored 0-6 with a minimum score of 0 and a maximum of 60. A higher score indicates greater symptomology.
psychotic symptomology | Change at 6 months
  Compass-10. The Compass-10 is a self-report scale that measures multiple symptoms associated with psychosis, including mood symptoms. It consists of 10-items, each scored 0-6 with a minimum score of 0 and a maximum of 60. A higher score indicates greater symptomology.
psychotic symptomology | Change at 4 months
  Compass-10. The Compass-10 is a self-report scale that measures multiple symptoms associated with psychosis, including mood symptoms. It consists of 10-items, each scored 0-6 with a minimum score of 0 and a maximum of 60. A higher score indicates greater symptomology.
psychotic symptomology | Change at 8 months
  modified-Colorado Symptom Index. The modified-Colorado Symptom Index is a 14-item, clinician-rated scale with items ranked 0-4. Total minimum score = 0. Total maximum score = 56. A higher score indicates greater symptomology.
psychotic symptomology | Change at 6 months
  modified-Colorado Symptom Index. The modified-Colorado Symptom Index is a 14-item, clinician-rated scale with items ranked 0-4. Total minimum score = 0. Total maximum score = 56. A higher score indicates greater symptomology.
psychotic symptomology | Change at 4 months
  modified-Colorado Symptom Index. The modified-Colorado Symptom Index is a 14-item, clinician-rated scale with items ranked 0-4. Total minimum score = 0. Total maximum score = 56. A higher score indicates greater symptomology.
depression | Change at 8 months
  abbreviated version of the Beck Depression Inventory-II (BDI-II) that has been previously validated (scale, min=0, max=21, higher mean score indicates more severe depressive symptomology)
depression | Change at 6 months
  abbreviated version of the Beck Depression Inventory-II (BDI-II) that has been previously validated (scale, min=0, max=21, higher mean score indicates more severe depressive symptomology)
depression | Change at 4 months
  abbreviated version of the Beck Depression Inventory-II (BDI-II) that has been previously validated (scale, min=0, max=21, higher mean score indicates more severe depressive symptomology)
quality of life | Change at 8 months
  4-item version of the Lehman Quality of Life Scale (min = 4, max =28, higher score is improved quality of life)
quality of life | Change at 6 months
  4-item version of the Lehman Quality of Life Scale (min = 4, max =28, higher score is improved quality of life)
quality of life | Change at 4 months
  4-item version of the Lehman Quality of Life Scale (min = 4, max =28, higher score is improved quality of life)
recovery | Change at 8 months
  5-item version of the Questionnaire about the Process of Recovery (scale, min=5, max=25, higher mean indicates more perceived recovery)
recovery | Change at 6 months
  5-item version of the Questionnaire about the Process of Recovery (scale, min=5, max=25, higher mean indicates more perceived recovery)
recovery | Change at 4 months
  5-item version of the Questionnaire about the Process of Recovery (scale, min=5, max=25, higher mean indicates more perceived recovery)
treatment motivation (intrinsic versus extrinsic) | Change at 8 months
  Treatment Motivation Questionnaire-Revised (TMQ-R). The Treatment Motivation Questionnaire-Revised is a 25-item self-assessment survey that assesses several elements of treatment motivation, each ranked 1-5. It is not a single scale that results in an overall score. Some items suggest greatest motivation at a 5 and least at a 1, but others suggest greatest motivation at a 1 and least at a 5.
treatment motivation (intrinsic versus extrinsic) | Change at 6 months
  Treatment Motivation Questionnaire-Revised (TMQ-R). The Treatment Motivation Questionnaire-Revised is a 25-item self-assessment survey that assesses several elements of treatment motivation, each ranked 1-5. It is not a single scale that results in an overall score. Some items suggest greatest motivation at a 5 and least at a 1, but others suggest greatest motivation at a 1 and least at a 5.
treatment motivation (intrinsic versus extrinsic) | Change at 4 months
  Treatment Motivation Questionnaire-Revised (TMQ-R). The Treatment Motivation Questionnaire-Revised is a 25-item self-assessment survey that assesses several elements of treatment motivation, each ranked 1-5. It is not a single scale that results in an overall score. Some items suggest greatest motivation at a 5 and least at a 1, but others suggest greatest motivation at a 1 and least at a 5.
Perceived coercion | Change at 8 months
  Modified version of the MacArthur Admission Experience Survey (AES). The MacArthur AES was developed as a self-assessment for assessing coercion and pressure during inpatient admission. It was previously modified for assisted outpatient treatment. We have modified it further to a 13-item scale for outpatient treatment generally. Each item is assessed as true or false, where true suggests great perception of pressure or coercion on some items, but less on others.
Perceived coercion | Change at 6 months
  Modified version of the MacArthur Admission Experience Survey (AES). The MacArthur AES was developed as a self-assessment for assessing coercion and pressure during inpatient admission. It was previously modified for assisted outpatient treatment. We have modified it further to a 13-item scale for outpatient treatment generally. Each item is assessed as true or false, where true suggests great perception of pressure or coercion on some items, but less on others.
Perceived coercion | Change at 4 months
  Modified version of the MacArthur Admission Experience Survey (AES). The MacArthur AES was developed as a self-assessment for assessing coercion and pressure during inpatient admission. It was previously modified for assisted outpatient treatment. We have modified it further to a 13-item scale for outpatient treatment generally. Each item is assessed as true or false, where true suggests great perception of pressure or coercion on some items, but less on others.
attendance rate | Change over 8 months
  number of appointments attended in a given period divided by number of appointments scheduled
attendance rate | Change at 6 months
  number of appointments attended in a given period divided by number of appointments scheduled
attendance rate | Change at 4 months
  number of appointments attended in a given period divided by number of appointments scheduled

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of North Carolina at Chapel Hill (ENCOMPASS Program), Raleigh, North Carolina
  - PEACE Program, Horizon House, Inc., Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadephia, Pennsylvania